CLINICAL TRIAL: NCT07204613
Title: The Effect of Aquatic Stimulation on the Development of Infants in the First Year of Life: A Pilot Study of a Randomized Controlled Clinical Trial
Brief Title: Infant Development and Early Aquatic Stimulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 68410223.3.0000.5108
Record Dates: First submitted 2025-08-29; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Infant Health; Child Development
Keywords: Aquatic Therapy; Child Development
MeSH Terms: interventions — Child Development

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Aquatic Stimulation (Experimental): Aquatic stimulation for babies up to one year of age, involving activities supervised by trained monitors, which aim to stimulate motor, cognitive, language and social development.
  Interventions: Behavioral: Aquatic stimulation for child development
- Control Group: Waiting List (No Intervention): The control group will consist of children who will remain on the waiting list to actively participate in aquatic stimulation after the research period.

INTERVENTIONS:
Behavioral: Aquatic stimulation for child development — The intervention will be conducted in a heated pool located in the Physiotherapy building of the Federal University of Jequitinhonha and Mucuri Valleys, Diamantina, Minas Gerais, Brazil. A total of 24 twice-weekly, 45-minute aquatic stimulation sessions will be offered over a 13-week intervention period. The sessions will follow a previously tested and refined aquatic stimulation protocol for infants. The experimental group will consist of 15 dyads (infant + parent or guardian) and three supervisors. Two will be inside the pool offering support and encouragement to parents and infants, and one will be outside the pool providing overall supervision of the children and controlling the time of each activity. The activities included in the aquatic intervention plan involve stimulation of expressive language, cognitive development, gross motor skills, fine motor skills, and social interaction.
  Arms: Experimental Group: Aquatic Stimulation

SUMMARY:
The objective of this study is to assess the feasibility of an aquatic stimulation protocol for infants up to one year of age. The main questions to be answered are:

Is the aquatic stimulation program, which involves recruitment, intervention, and reassessment, feasible and feasible on a larger scale? Was the aquatic stimulation protocol able to promote improvements in child development compared to the control group?

Researchers will compare the intervention group with a control group, which will be included on the waiting list, to determine whether aquatic stimulation promotes improved child development.

Eligible participants will be assessed, and then a random selection will be made by an independent researcher to determine the control and experimental groups. The experimental group will receive aquatic stimulation through a group class, with activities that stimulate language, cognitive, fine and gross motor skills, as well as social interaction. The control group will remain on the waiting list throughout the intervention. Monthly messages will be sent to both groups to collect information about the infant's health. Interventions will occur twice a week for 45 minutes over a three-month period. Immediately afterward, the children and their parents/guardians will be reevaluated. Children in the control group will be guaranteed a spot to receive aquatic stimulation after the intervention period. The data will be tabulated, analyzed, and subsequently published scientifically.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 months to 7 months and 29 days with expressed interest from their parents and/or guardians in participating in the outreach project "Nada Melhor: Aquatic Stimulation for Babies";
* Participation in the research with authorization and consent from their parents or guardians.
* Availability to attend aquatic stimulation classes on previously defined days and times (Tuesdays and Thursdays, 6:00 PM to 7:00 PM).

Exclusion Criteria:

* Children with neurological disorders such as cerebral palsy or syndromes affecting cognitive, linguistic, and motor skills, mental or psychiatric disorders, and autism;
* Children with prior experience in an aquatic environment under the supervision of a professional.

Ages: 3 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Intervention Protocol | 4 months
  Measure Unit: Composite Score (0-100)
  Description: A single feasibility score will be calculated by aggregating multiple indicators: number of sessions attended/missed, dropout rate, impact of inclusion/exclusion criteria on recruitment, rate of adverse events, parental satisfaction, and adherence to protocol activities. Each indicator will be scored and combined into a composite score ranging from 0 (lowest feasibility) to 100 (highest feasibility), reflecting the overall feasibility of the intervention protocol.
Child Development | From registration to end of re-evaluation = 5 months
  Child development will be assessed using the Bayley-III instrument. The assessment begins with age-appropriate tasks and is scored as 1 if the task is completed and 0 if it is not. The assessment ends when the child fails five consecutive tasks. Each domain generates a raw score, which can be converted into balanced and composite scores using tables provided in the manual. The balanced score will classify the child from 1 to 19. The mean is 10 and a standard deviation of ±3 points, being classified as expected (7 to 13 points), below expected (<7 points), and above expected (<13 points). The composite score is based on age norms, classifying the child from 40 to 160. The mean score is 100, with a standard deviation of ±15 points.

SECONDARY OUTCOMES:
Socioeconomic classification of the family | 4 months
  For economic classification, the Brazilian Economic Classification Criteria (CCEB) from the Brazilian Association of Research Companies (ABEP) 2018 will be used. This criteria assigns a score based on the assets and education of the head of the household. Based on this score, the family is classified on an ordinal scale from E to A.
Opportunity for motor stimulation at home | 4 months
  The Affordances in the Home Environment for Motor Development (AHEMD) will be used to assess the opportunities children have at home. The instrument has been translated and validated for the Brazilian population and aims to assess the quality and quantity of opportunities for motor stimulation in children's homes. The instrument should be completed based on reports from parents or caregivers. It is divided into two categories, according to the child's age: 2 to 18 months and 18 to 42 months. After completing the questionnaire, the scores for each dimension are calculated by adding the points from the questions and then totaled to obtain the total score. The maximum score for the questionnaire is 20 points, and it can be classified as high (17 to 20 points), medium (10 to 16 points), and low (less than 9 points).
Global Development and Child Behavior | 4 months
  To assess overall development, we used an instrument translated and adapted to the Brazilian version of the "Survey of Well-being of Young Children (SWYC)." This instrument is presented in the form of a compilation of questionnaires, 12 in total, in which each section assesses a domain of the child's well-being, and a score is generated at the end of each domain. Based on this score and the child's age, the administrator can use a table to determine whether the score is the minimum expected for that age. The SWYC can be accessed at: https://www.tuftsmedicine.org/medical-professionals-trainees/academic departments/department-pediatrics/survey-well-being-young-children/age-specific-forms.
Sociodemographic and biological factors that can influence child development | 1 day
  Initially, parents and/or guardians will answer a questionnaire prepared by the authors about sociodemographic and biological data characterizing the sample, such as: sex, age, aspects related to the gestational period, family history, and data on the infant's health and habits.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal dos Vales do Jequitinhonha e Mucuri, Diamantina, Minas Gerais, Brazil